CLINICAL TRIAL: NCT05799040
Title: Evaluation of the Effectiveness of the Self-developed Pulmonary Lobar Ventilation Detector
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: 2022-NHLHCRF-LX-01-0202-3
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Self-developed pulmonary lobar ventilation detector
  Interventions: Device: Self-developed pulmonary lobar ventilation detector
- imported Chartis detection system
  Interventions: Device: Chartis detection system

INTERVENTIONS:
Device: Self-developed pulmonary lobar ventilation detector — The participants would evaluated by the self-developed pulmonary lobar ventilation detector.
  Groups: Self-developed pulmonary lobar ventilation detector
Device: Chartis detection system — The participants would evaluated by the Chartis detection system.
  Groups: imported Chartis detection system

SUMMARY:
The goal of observational study is to Evaluation of the effectiveness of the self-developed pulmonary lobar ventilation detector in Chronic Obstructive Pulmonary Disease. The main question it aims to answer are:Evaluation of the effectiveness of the self-developed pulmonary lobar ventilation detector.

Participants will use the self-developed pulmonary lobar ventilation detector and the imported Chartis detection system to evaluate the target pulmonary lobar collateral ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease who meet the GOLD diagnostic criteria
* FEV1 ≤ 45% pred and FEV1/FVC<70%
* TLC>100% pred and RV>175% pred
* CAT≥18
* >50% of emphysema destruction
* Smoking prohibition>6 months
* Sign the informed consent form

Exclusion Criteria:

* PaCO2>8.0 kPa, or PaO2<6.0 kPa
* 6-minute walking test<160m
* Obvious chronic bronchitis, bronchiectasis or other infectious lung diseases
* Three hospitalizations due to pulmonary infection in the past 12 months before the baseline assessment
* Previous lobectomy, LVRS or lung transplantation
* LVEF<45% and or RVSP>50mmHg
* Anticoagulant therapy that cannot be stopped before surgery
* The patient has obvious immune deficiency
* Participated in other lung drug studies within 30 days before this study
* Pulmonary nodules requiring intervention
* Any disease or condition that interferes with the completion of the initial or subsequent assessment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect of lung volume reduction surgery | 1 month after bronchoscopic valve lung volume reduction
  Lung CT
Therapeutic effect of lung volume reduction surgery | 3 months after bronchoscopic valve lung volume reduction
  Lung CT
Therapeutic effect of lung volume reduction surgery | 6 months after bronchoscopic valve lung volume reduction
  Lung CT
the integrity of interlobar fissure | Before bronchoscopic valve lung volume reduction
  Use the self-developed pulmonary lobar ventilation detector and the imported Chartis detection system to evaluate the target pulmonary lobar collateral ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China